CLINICAL TRIAL: NCT01092130
Title: An Open-label, Blinded-endpoint, Randomized, Prospective Trial Investigating the Effects of Vitamin D Administration on Plasma Renin Activity in Patients With Stable Chronic Heart Failure
Brief Title: Study to Investigate the Effects of Vitamin D Administration on Plasma Renin Activity in Patients With Stable Chronic Heart Failure
Acronym: VitD-CHF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Netherlands Foundation for Cardiovascular Excellence (Unknown)
Responsible Party: Principal Investigator, Willem-Peter Theodoor Ruifrok, MD, PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WTR-ECG-4
Record Dates: First submitted 2010-03-12; First posted 2010-03-24 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Heart Failure
Keywords: Heart failure; Vitamin D; Plasma renin activity; Renin angiotensin system
MeSH Terms: conditions — Heart Failure | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin D (Experimental): Patients were randomized by an automated computer system to 2000 IU oral cholecalciferol once daily or control (i.e. no extra medication), in a 1:1 ratio for a period of six weeks. Blood was collected in a sitting position on visits 2-4 and patients were asked to collect 24h urine samples prior to visits 2 and 4. Heart failure medication was maintained unchanged throughout the trial. Changes in diuretic dose were permitted if necessary to treat decompensation or renal dysfunction.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — 2000 IU vitamin D daily, for 6 weeks
  Other Names: Colecalciferol

SUMMARY:
The renin-angiotensin system (RAS) is a regulatory system that plays an essential role in patients with chronic heart failure (CHF). Plasma renin activity (PRA) is a strong and independent predictor of outcome, also in the presence of ACE inhibitors (ACE-i) and/or angiotensin receptor blockers (ARBs). Recently, it has been shown that vitamin D regulates renin transcription by activating the vitamin D receptor (VDR). Thus, specific activation of the VDR represents a novel target for therapeutic intervention in CHF. Currently, clinical data are lacking. The investigators aim to investigate the effect of the administration of vitamin D in patients with CHF.

ELIGIBILITY:
Inclusion Criteria:

* Out clinical patients ≥ 18 years of age, male or female.
* Patients with a diagnosis of chronic heart failure (NYHA Class II, III or IV).
* Patients must at least be treated with an ACE-i at a stable dose (at least enalapril 10 mg daily or any other ACE-i, e.g. ramipril, quinapril, lisinopril, fosinopril, perindopril, trandolapril; on equivalent doses, or maximum tolerated dose) or if intolerant to ACE-i with ARB therapy (Candesartan 8 mg daily or any other ARB in equivalent dose, or maximum tolerated dose) for at least 4 weeks prior to visit 1.
* Patients must be treated with a beta blocker unless contraindicated or not tolerated at a stable dose for at least 4 weeks prior to visit 1 (for patients not on target dose or in absence of that medication, the reason should be documented).
* Concomitant use of ACE-i and/or ARB and/or aldosterone antagonist is permitted.

Exclusion Criteria:

* LVEF >45% at visit 1 (local measurement, measured within the past 12 months assessed by echocardiogram, MUGA or ventricular angiography).
* History of hypersensitivity to the study drugs.
* Patients with phenylketonuria.
* Patients with fructose intolerance.
* Current acute decompensated heart failure.
* Hypercalcemia (>2.65 mmol/l, corrected for albumin).
* Hypercalciuria.
* Estimated glomerular filtration fraction (eGFR) between 30 and 60 ml/min/1.73m2 as measured by the modified of diet in renal disease (MDRD) formula.
* Nephrolithiasis.
* Sarcoidosis.
* Use of the following medication: corticosteroids, thyroxin, anti epileptic drugs, tetracyclines, quinolones
* Intake of supplements containing vitamin D and/or calcium.
* Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or major vascular surgery, percutaneous coronary intervention (PCI) or carotid angioplasty, within the past 3 months.
* Coronary or carotid artery disease likely to require surgical or PCI.
* Right heart failure due to severe pulmonary disease.
* Diagnosis of peripartum or chemotherapy induced cardiomyopathy within the last year.
* Patients with a history of heart transplant or who are on a transplant list or with LVAD device (left ventricular assistance device).
* Documented ventricular arrhythmia with syncopal episodes within past 3 months that is untreated.
* Documented history of ventricular tachycardia or ventricular fibrillation without ICD (internal cardiac defibrillator).
* Symptomatic bradycardia, or second or third degree heart block without a pacemaker.
* Implantation of a CRT (cardiac resynchronization therapy) device within prior 3 months.
* Presence of hemodynamically significant mitral and /or aortic valve disease, except mitral regurgitation secondary to left ventricular dilatation.
* Presence of hemodynamically significant obstructive lesions of left ventricular outflow tract, including aortic stenosis.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs.
* Any history of pancreatic injury, pancreatitis or evidence of impaired pancreatic function/injury as indicated by abnormal lipase or amylase.
* Primary liver disease considered to be life threatening.
* Currently active gastritis, duodenal or gastric ulcers, or gastrointestinal/rectal bleeding during the 3 months prior to Visit 1.
* History or presence of any other diseases (i.e. including malignancies) with a life expectancy of < 5 years.
* Current double-blind treatment in heart failure (HF) trials.
* Participation in an investigational drug study at the time of enrollment or within the past 30 days or 5 half lives of enrollment whichever is longer.
* Any surgical or medical condition that in the opinion of the investigator or medical monitor would jeopardize the evaluation of efficacy or safety.
* History of noncompliance to medical regimens and patients who are considered potentially unreliable.
* Pregnant or lactating women.
* Treatment with any of the following drugs within the past 4 weeks prior to Visit 1 (T0):
* Direct renin inhibition including Aliskiren
* Intravenous vasodilator and/or inotropic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Plasma Renin Activity | 6 weeks
  The primary endpoint of this study is the PRA after 6 weeks of treatment with vitamin D compared to the PRA after 6 weeks without treatment.

SECONDARY OUTCOMES:
Safety endpoints are biochemical indices of kidney function and bone homeostasis | 6 weeks
To evaluate the effect of vitamin D administration on plasma values of additional markers of renin-angiotensin system activity, including angiotensin II, angiotensin converting enzyme activity and chymase activity | 6 weeks
To evaluate the effect of vitamin D administration on different markers of the vitamin D cascade, such as vitamin D, calcium, phosphate and PTH (parathyroid hormone) | 6 weeks
To evaluate the effect of vitamin D administration on plasma levels of NT-proBNP | 6 weeks
To evaluate the effect of vitamin D administration on urinary levels of markers of glomerular and tubular damage | 6 weeks
To evaluate the effect of vitamin D administration on extracellular matrix markers (PIIINP, PICP, PINP) and degradation markers (MMP1, MMP9, TIMP1, MMP1/TIMP1-complex) | 6 weeks
To evaluate the effect of vitamin D administration on NYHA-class | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: W. T. Ruifrok, MD, Principal Investigator — University Medical Center Groningen; R. A. de Boer, MD, PhD, Study Director — University Medical Center Groningen; W. H. van Gilst, PhD, Study Chair — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Schroten NF, Ruifrok WP, Kleijn L, Dokter MM, Sillje HH, Lambers Heerspink HJ, Bakker SJ, Kema IP, van Gilst WH, van Veldhuisen DJ, Hillege HL, de Boer RA. Short-term vitamin D3 supplementation lowers plasma renin activity in patients with stable chronic heart failure: an open-label, blinded end point, randomized prospective trial (VitD-CHF trial). Am Heart J. 2013 Aug;166(2):357-364.e2. doi: 10.1016/j.ahj.2013.05.009. Epub 2013 Jun 24. PMID 23895820